CLINICAL TRIAL: NCT05573646
Title: Online Group-based Dual-task Training to Improve Cognitive Function of Community-dwelling Older Adults: A Feasibility Study
Brief Title: Online Group-based Dual-task Training to Improve Cognitive Function of Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Dr. Pui-Hing Chau, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19200991
Record Dates: First submitted 2022-09-25; First posted 2022-10-10 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Aging Well

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-task training (Experimental): Dual-task training group
  Interventions: Other: Dual-task training
- Attention control (Other): Attention control group
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: Dual-task training — Participants will receive a one-hour online group-based dual-task training session twice a week for 12 weeks, giving a total intervention time of 24 hours. A co-design approach will be adopted to develop the training components in the dual-tasks. For the cognitive training component, arithmetic operation, verbal fluency, and upper limb/ finger movements are included. For the physical training component, we select chair-based exercises are included. A group-based training mode led by a facilitator will be adopted. During the session, participants will be asked to turn on their camera so that they can see and interact with each other. They will also have their audio on as they will have to participate in the cognitive tasks by voicing out their answers.
  Arms: Dual-task training
Other: Attention Control — Participants will receive eight one-hour online group-based interactive education on health topics other than exercise and cognitive health.
  Arms: Attention control

SUMMARY:
Objectives: This study aims to explore the feasibility, acceptance, and efficacy of online group-based dual-task training as an intervention for improving cognitive function among community-dwelling older adults.

Hypothesis to be tested: We hypothesize that after the intervention, there will be an improvement in the participants' cognitive function as compared with pre-intervention status and with the control group. Also, lower-limb muscle strength and psychosocial wellbeing will be improved after the intervention.

Design and subjects: This is a randomised controlled feasibility study. The target population is community-dwelling older adults with access to an online meeting platform. About 75 participants will be recruited and randomised to the intervention and attention control groups in a ratio of 2:1. Intervention group will receive 60 minutes of online group-based dual-task training twice a week for 12 weeks led by a trained facilitator. Cognitive training components include arithmetic operation, verbal fluency, and upper limb/finger movement. Physical training components are chair-based exercises. The training components will be selected using a co-design approach.

Instruments: Memory Inventory in Chinese (MIC), Digit Span Test, Victoria Stroop Test, Montreal Cognitive Assessment 5-Minutes (Hong Kong Version).

Main outcome measures: Subjective memory complaints as measured by MIC.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years and above,
* no communication problems,
* able to communicate in Chinese, and
* able to use an online meeting platform.

Exclusion Criteria:

* contraindications to chair-based exercises, and
* engagement in any kind of cognitive training three months prior to the study or during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline subjective memory complaints at 6 weeks | Six weeks after baseline
  Measured by Memory Inventory in Chinese. The sum of score ranges from 0 to 108, higher score indicates more memory complaints.
Change from baseline subjective memory complaints at 12 weeks | 12 weeks after baseline
  Measured by Memory Inventory in Chinese. The sum of score ranges from 0 to 108, higher score indicates more memory complaints.
Change from baseline subjective memory complaints at 18 weeks | 18 weeks after baseline
  Measured by Memory Inventory in Chinese. The sum of score ranges from 0 to 108, higher score indicates more memory complaints.

SECONDARY OUTCOMES:
Change from baseline cognitive status at 6 weeks | Six weeks after baseline
  Measured by the Montreal Cognitive Assessment 5-Minutes (Hong Kong Version) (HK-MoCA 5-Min) protocol. The total score ranges from 0 to 30; a higher score indicates better cognitive status.
Change from baseline cognitive status at 12 weeks | 12 weeks after baseline
  Measured by the Montreal Cognitive Assessment 5-Minutes (Hong Kong Version) (HK-MoCA 5-Min) protocol. The total score ranges from 0 to 30; a higher score indicates better cognitive status.
Change from baseline cognitive status at 18 weeks | 18 weeks after baseline
  Measured by the Montreal Cognitive Assessment 5-Minutes (Hong Kong Version) (HK-MoCA 5-Min) protocol. The total score ranges from 0 to 30; a higher score indicates better cognitive status.
Change from baseline working memory at 6 weeks | Six weeks after baseline
  Measured by Digit Span Test. The longer the series, the better the condition.
Change from baseline working memory at 12 weeks | 12 weeks after baseline
  Measured by Digit Span Test. The longer the series, the better the condition.
Change from baseline working memory at 18 weeks | 18 weeks after baseline
  Measured by Digit Span Test. The longer the series, the better the condition.
Change from baseline executive function at 6 weeks | Six weeks after baseline
  Measured by Chinese version of the Victoria Stroop Test, with more time and errors as worse condition.
Change from baseline executive function at 12 weeks | 12 weeks after baseline
  Measured by Chinese version of the Victoria Stroop Test, with more time and errors as worse condition.
Change from baseline executive function at 18 weeks | 18 weeks after baseline
  Measured by Chinese version of the Victoria Stroop Test, with more time and errors as worse condition.
Change from baseline lower-limb muscle strength at 6 weeks | Six weeks after baseline
  Measured by the 5-times chair stand task. The longer the time participants use to finish the task, the poorer the performance.
Change from baseline lower-limb muscle strength at 12 weeks | 12 weeks after baseline
  Measured by the 5-times chair stand task. The longer the time participants use to finish the task, the poorer the performance.
Change from baseline lower-limb muscle strength at 18 weeks | 18 weeks after baseline
  Measured by the 5-times chair stand task. The longer the time participants use to finish the task, the poorer the performance.
Change from baseline happiness at 6 weeks | Six weeks after baseline
  Measured by the Chinese version of the 4-item Subjective Happiness Scale. The score is the average of the four items, and ranges from 1 to 7; a higher score indicates a higher happiness level.
Change from baseline happiness at 12 weeks | 12 weeks after baseline
  Measured by the Chinese version of the 4-item Subjective Happiness Scale. The score is the average of the four items, and ranges from 1 to 7; a higher score indicates a higher happiness level.
Change from baseline happiness at 18 weeks | 18 weeks after baseline
  Measured by the Chinese version of the 4-item Subjective Happiness Scale. The score is the average of the four items, and ranges from 1 to 7; a higher score indicates a higher happiness level.
Change from baseline depressive symptoms at 6 weeks | Six weeks after baseline
  Measured by the Patient Health Questionnaire-9. The scale ranged from 0 to 27, higher score indicates higher level of depressive symptoms.
Change from baseline depressive symptoms at 12 weeks | 12 weeks after baseline
  Measured by the Patient Health Questionnaire-9. The scale ranged from 0 to 27, higher score indicates higher level of depressive symptoms.
Change from baseline depressive symptoms at 18 weeks | 18 weeks after baseline
  Measured by the Patient Health Questionnaire-9. The scale ranged from 0 to 27, higher score indicates higher level of depressive symptoms.
Change from baseline social isolation/integration at 6 weeks | Six weeks after baseline
  Measured by the Chinese version of the 6-item Lubben Social Network Scale. The total score ranges from 0 to 30; a higher score indicates a better social network.
Change from baseline social isolation/integration at 12 weeks | 12 weeks after baseline
  Measured by the Chinese version of the 6-item Lubben Social Network Scale. The total score ranges from 0 to 30; a higher score indicates a better social network.
Change from baseline social isolation/integration at 18 weeks | 18 weeks after baseline
  Measured by the Chinese version of the 6-item Lubben Social Network Scale. The total score ranges from 0 to 30; a higher score indicates a better social network.
Change from baseline instrumental activity of daily living at 6 weeks | Six weeks after baseline
  Measured by Lawton's eight selected tasks. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Change from baseline instrumental activity of daily living at 12 weeks | 12 weeks after baseline
  Measured by Lawton's eight selected tasks. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Change from baseline instrumental activity of daily living at 18 weeks | 18 weeks after baseline
  Measured by Lawton's eight selected tasks. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Hing Chau, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- Nursing Home, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chau PH, Cheung DST, Kwok JYY, Chan WC, Yu DSF. Online Group-Based Dual-Task Training to Improve Cognitive Function of Community-Dwelling Older Adults: Randomized Controlled Feasibility Study. JMIR Aging. 2025 May 16;8:e67267. doi: 10.2196/67267. PMID 40378407